CLINICAL TRIAL: NCT02745639
Title: Preoperative Chemoradiation With VMAT-SIB in Rectal Cancer: a Phase II Study.
Brief Title: Preoperative Chemoradiation With VMAT-SIB in Rectal Cancer
Acronym: GRACE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Lorenzo Fuccio, Associate professor of Gastroenterology, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GRACE-RECTUM-1
Record Dates: First submitted 2016-04-17; First posted 2016-04-20 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Rectal Neoplasms
Keywords: rectal cancer; radiotherapy; chemotherapy; VMAT; toxicity
MeSH Terms: conditions — Rectal Neoplasms | interventions — XELOX; Oxaliplatin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- VMAT-SIB + XELOX (Experimental): A VMAT-SIB technique was used. Radiation dose prescribed to PTV2 was 45 Gy (1.8 Gy/fraction), five sessions weekly in 25 daily fractions. A simultaneous boost was delivered on PTV1 with a total dose of 57.5 Gy (2.3 Gy/fraction). Dose-volume histograms (DVHs) were calculated for the PTV1, PTV2 and Organs at risks.
  The prescribed concurrent chemotherapy consisted of oxaliplatin infusion 130 mg/m2 on days 1, 17, 35 and capecitabine 1650 mg/m2 daily (825 mg/m² twice daily, 5 days/week) over all the treatment.
  Interventions: Radiation: VMAT-SIB; Drug: XELOX

INTERVENTIONS:
Radiation: VMAT-SIB — Radiation dose prescribed to PTV2 was 45 Gy (1.8 Gy/fraction), five sessions weekly in 25 daily fractions. A simultaneous boost was delivered on PTV1 with a total dose of 57.5 Gy (2.3 Gy/fraction). Dose-volume histograms (DVHs) were calculated for the PTV1, PTV2 and OARs. Patients were treated only if the relative variations of the bone markers between the images were within 3 mm along the three spatial directions. Planning and delivery processes underwent to systematic independent-check procedures.
Drug: XELOX — The prescribed concurrent chemotherapy consisted of oxaliplatin infusion 130 mg/m2 on days 1, 17, 35 and capecitabine 1650 mg/m2 daily (825 mg/m² twice daily, 5 days/week) over all the treatment. An adequate blood count was necessary to start each chemotherapy infusion. Adjuvant chemotherapy was recommended on patients with high risk factors at pathological examination and decision was left to medical oncologists discretion.
  Other Names: Oxaliplatin + Capecitabine

SUMMARY:
This was a prospective phase II study on patients with locally advanced rectal cancer or local recurrence, to evaluate the pathological response and resectability of a neoadjuvant treatment based on the use of a combined treatment with VMAT-SIB and two drugs chemotherapy ( XELOX).

DETAILED DESCRIPTION:
This was a prospective phase II study on patients with LARC or local recurrence, to evaluate the pathological response and resectability of a neoadjuvant treatment based on the use of a combined treatment with VMAT-SIB and two drugs chemotherapy ( XELOX).

The primary aim was to asses the pathological response rate. Key secondary aim was the acute toxicity. Secondary aims were local control, disease-free survival (DFS) and overall survival (OS).

The follow-up period of each subjects started at the end of combined treatment and concluded after a period of maximum 60 months or until death.

ELIGIBILITY:
Inclusion Criteria: i) histologically proven rectal adenocarcinoma (cT3-4N0-2 or cT2N1-2 or locally recurrent) beginning within 12 cm from the anal verge; ii) age ≥ 18 years; iii) Eastern Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.

Exclusion Criteria: i) history of chemotherapy and/or pelvic radiotherapy; ii) previous treatment with immunotherapy; iii) metastatic patient; iv) presence of active intestinal inflammation or uncontrolled pelvic inflammation; v) pregnant and/or breastfeeding patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2010-02; Primary Completion 2013-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Pathological response rate | 6-8 weeks after chemoradiotherapy
  Pathological response was determined according to the TNM classification system of the American Joint Committee on Cancer. The complete resection of the tumor (R) with no histological proven residual disease in the surgical specimen, was defined as pathological complete response (pCR =pT0). Near complete response (pTmic) was defined as the presence of a number of neoplastic cells inferior to 10%.

SECONDARY OUTCOMES:
Acute Toxicity | During radiation treatment and at the first follow-up visit (4 weeks after RT).
  To score acute toxicity CTCAE v.3.0 was used

CONTACTS AND LOCATIONS:
Overall Officials: Alessio G Morganti, Professor, Study Director — Division of Radiation Oncology, S.Orsola-Malpighi Hospital, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Yes
International Journals